CLINICAL TRIAL: NCT05223764
Title: Why Are They Not Coming Back? A Single-center Follow-up Study in Fertility Preservation in Oncological Women.
Brief Title: Why Are Fertility Preservation Patients Not Coming Back?
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 72/20
Record Dates: First submitted 2022-01-24; First posted 2022-02-04 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-01

CONDITIONS: Fertility Issues; Cancer
MeSH Terms: conditions — Infertility; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fertility preservation population: all women who underwent oocyte cryopreservation cycles for oncological purposes from January 2001 to December 2017 at Fertility Center of Humanitas Research Hospital, Rozzano (Milano), Italy
  Interventions: Other: Follow up survey

INTERVENTIONS:
Other: Follow up survey — phone call follow-up to investigate women's decision not to return for embryo transfer after cancer treatment.

SUMMARY:
This is a single-center retrospective study carried out with a phone call follow-up to investigate women's decision not to return for criopreserved ovocytes use after cancer treatment. The study database includes all women who underwent fertility preservation cycles at a third-level university-affiliated center from January 2001 to December 2017.

Patients were asked a set of standardized questions whose purpose was to investigate their present health conditions, cancer treatment and any potential relapses, their family projects and sentimental status, any spontaneous conception, and why they had not yet returned for embryo transfer.

All data were recorded anonymously in our dataset.

DETAILED DESCRIPTION:
All women who underwent oocyte cryopreservation cycles for oncological purposes from January 2001 to December 2017 at Fertility Center of Humanitas Research Hospital, Rozzano (Milano), Italy, were contacted.

The survey's purpose was to investigate their present health conditions, cancer treatment and any potential relapses, their family projects and sentimental status, any spontaneous conception, and why they had not yet returned for oocytes use.

ELIGIBILITY:
Inclusion Criteria:

The study database includes all women who underwent fertility preservation cycles at a third-level university-affiliated center

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Women with an oncological diagnosis who underwent ovarian stimulation and oocytes retrivial and cryopreservation for fertility preservation
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
return rate | from January 2001 to December 2021
  return rate of cancer patients who underwent fertility preservation

CONTACTS AND LOCATIONS:
Locations (1):
- Valentina Immediata, Milan, MI, Italy

REFERENCES:
- [Derived] Immediata V, Cirillo F, Baggiani A, Zanagnolo MF, Ronchetti C, Morenghi E, Cesana A, Specchia C, Levi-Setti PE. Why are they not coming back? A single-center follow-up study on oncological women oocyte's storing for fertility preservation. Front Endocrinol (Lausanne). 2022 Dec 6;13:1054123. doi: 10.3389/fendo.2022.1054123. eCollection 2022. PMID 36561560